CLINICAL TRIAL: NCT03533023
Title: Optimizing Circadian Rhythms by Regulating Eating Patterns to Reduce Cardiometabolic Disease Risk Among Firefighters--The Healthy Heroes Study
Brief Title: The Healthy Heroes Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Salk Institute for Biological Studies (Other)
Responsible Party: Principal Investigator, Pam Taub, MD, Associate Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 172083
Record Dates: First submitted 2018-04-19; First posted 2018-05-22 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Shift Workers' Health; Time Restricted Eating; Fasting
Keywords: Firefighters; San Diego Fire and Rescue; Cardiometabolic Health; First Responder; Shift Workers; Time-Restricted Eating; Fasting
MeSH Terms: conditions — Intermittent Fasting; Fasting | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRE + SOC (Experimental): Time Restricted Eating + Standard of Care
  Interventions: Behavioral: Time Restricted Eating + Standard of Care
- SOC (Other): Standard of Care
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Time Restricted Eating + Standard of Care — Participants in this arm will adhere to a daily, consistent 10-hr eating window for the course of the study as well as receive nutritional counseling from the study dietician.
  Other Names: Time Restricted Eating
  Arms: TRE + SOC
Behavioral: Standard of Care — Participants in this arm will receive nutritional counseling from the study dietician, but will not be required to adopt a 10-hr eating window.
  Arms: SOC

SUMMARY:
This is the first study of its kind to assess and test an intervention to improve biological rhythms and general health of shift workers, specifically first responders with San Diego Fire and Rescue. In a randomized control trial, investigators intend to measure the health impact of Time Restricted Eating in emergency responders who work a 24-hour shift schedule.

DETAILED DESCRIPTION:
Participants will be randomly assigned to a control group of behavioral nutrition counseling (standard of care) or the intervention group of standard of care with the addition of adopting a 10 hour eating window for one year (TRE). For the first 3 months of intervention, participants will be monitored closely by the research team. For the following 9 months, participants will be in a self-monitored intervention period. Investigators will evaluate the impact of TRE on blood glucose levels, biomarkers, sleep/mood, and weight loss. These assessments will be made at baseline, at the end of the 12-week monitored intervention period, and every 3 months (months 6, 9, and 12) during the self-monitored intervention period for one year. Food/drink intake, activity, and sleep will be monitored with the smartphone myCircadianClock application ("mCC app") throughout the study. A continuous glucose monitor, a wrist-worn actigraphy device, and questionnaires will also be used during the study.

ELIGIBILITY:
As per recommendations from the fire department, fire department unions, and funding agencies, we did not require compromised health measures (e.g. hyperglycemia, hypertension, etc.) as inclusion criteria for they would be discriminatory against some firefighters.

Inclusion Criteria:

* Firefighter or work a 24-hr shift schedule with San Diego Fire and Rescue
* Age: 21-65 years
* Own a smartphone (Apple or Android Operating System)
* If participants are on cardiovascular medications (HMG-CoA reductase inhibitors (statins), other lipid modifying drugs (including over the counter drugs such as red yeast rice and fish oil), anti-hypertensive, anti-diabetes drugs), no dose adjustments will be allowed during the study period

Exclusion Criteria:

* Insulin-dependent diabetes mellitus
* Presence of acute chronic inflammatory or autoimmune disease (defined by acute symptoms or C-reactive protein >10 mg/L), malabsorption syndromes, liver disease, or kidney disease (stage 3 or greater)
* Uncontrolled thyroid disease
* Intake of drugs likely to interfere with study endpoints, including corticosteroids, anabolic steroids, anti-psychotics, antiretroviral drugs, and immunosuppressive drugs (within 3 months of starting the study)
* Presence or recent history of anemia (hematocrit <33% within 3 months of starting the study)
* History of bariatric surgery
* Pregnant or breast-feeding women
* Current or recent (within 12 months of starting the study) pregnancy or breastfeeding, or intention of becoming pregnant in the next 6 months
* Any cancer other than non-melanoma skin cancer in the last 3 years
* On a special or prescribed diet for other reasons (e.g. Celiac disease)
* Depression determined by the Beck Depression Inventory (BDI)
* Planned international travel during study period
* Insufficient logging on the mCC app (does not log at least 2 entries a day for 10 of 14 days) during baseline will exclude from being randomized into the intervention period

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the impact of TRE on glucose homeostasis at end of intervention compared to baseline | primary endpoint=12-week intervention (compared to 2-week baseline); follow-up will be at 1-year
  Measured by an ambulatory continuous glucose monitoring device and blood work throughout the study.
  Note: Significant changes expected in participants who had elevated glucose homeostasis at baseline. No significant changes expected in those within normal ranges at baseline. Primary endpoint analysis will be done by comparing baseline and 12-week intervention.
Assess the feasibility and adherence of TRE | primary endpoint=12-week intervention (compared to 2-week baseline); follow-up will be at 1-year
  Measured by percentage of days logged that participants ate within their 10-hour window and by end of study responses.
  Note: Significant changes expected in participants in the TRE arm of the study on and off shift. No significant changes expected in the standard of care arm of the study. Primary endpoint analysis will be done by comparing baseline and 12-week intervention.

SECONDARY OUTCOMES:
Assess changes in metabolic biomarkers in response to TRE at end of intervention compared to baseline | Timeframe: primary endpoint=12-week intervention (compared to 2-week baseline); follow-up will be at 1-year
  Measured with blood biochemistry.Measured with blood biochemistry under TRE, including, but not limited to: fasting glucose, HbA1c, cholesterol, and triglycerides.
  Note: Significant changes expected in participants who had abnormal levels at baseline (e.g. elevated LDL cholesterol, low HDL cholesterol, elevated triglycerides). No significant changes expected in those were within normal ranges at baseline.
Systolic blood pressure (mmHg) in response to TRE at end of intervention compared to baseline | Timeframe: primary endpoint=12-week intervention (compared to 2-week baseline); follow-up will be at 1-year
  Measured at baseline and during TRE intervention. Note: Significant changes expected in participants who had elevated systolic blood pressure at baseline. No significant changes expected in those without elevated systolic blood pressure at baseline.
Diastolic blood pressure (mmHg) in response to TRE at end of intervention compared to baseline | primary endpoint=12-week intervention (compared to 2-week baseline); follow-up will be at 1-year
  Measured at baseline and during TRE intervention. Note: Significant changes expected in participants who had elevated diastolic blood pressure at baseline. No significant changes expected in those without elevated diastolic blood pressure at baseline.
Body weight (kg) | primary endpoint=12-week intervention (compared to 2-week baseline); follow-up will be at 1-year
  Measured on a digital scale. Note: Significant changes expected in participants who had elevated weight at baseline. No significant changes expected in those who were not overweight at baseline.

OTHER OUTCOMES:
Body mass index (kg/m^2) | primary endpoint=12-week intervention (compared to 2-week baseline); follow-up will be at 1-year
  Calculated from body weight (kg) and height (m). Note: Significant changes expected in participants who had elevated BMI at baseline. No significant changes expected in those whose BMI was not elevated at baseline.
Waist and hip circumference (cm) | primary endpoint=12-week intervention (compared to 2-week baseline); follow-up will be at 1-year
  Measured with standardized body tape measure. Note: Significant changes expected in participants who had increased waist and hip circumference at baseline. No significant changes expected in those without increased waist and hip circumference at baseline.
Hip (cm)/waist (cm) ratio | primary endpoint=12-week intervention (compared to 2-week baseline); follow-up will be at 1-year
  Measured using tape measure. Note: Significant changes expected in participants who had an increased hip/waist ratio at baseline. No significant changes expected in those without increases at baseline
Body composition including but not limited to fat percentage (%), fat mass (kg), and lean mass (kg) | primary endpoint=12-week intervention (compared to 2-week baseline); follow-up will be at 1-year
  Measured by Tanita Digital Scale. Note: Significant changes expected in participants who had elevations levels at baseline. No significant changes expected in those without elevations at baseline.
Questionnaires (quality of life, sleep, and health) | primary endpoint=12-week intervention (compared to 2-week baseline); follow-up will be at 1-year
  Measured by SF-36, PSQI, and ESS. Note: Significant changes expected in participants who had decreased self-reporting of the above-mentioned questionnaires at baseline. No significant changes expected in those without decreases at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Pam Taub, MD, Principal Investigator — UCSD
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Derived] Manoogian ENC, Zadourian A, Lo HC, Gutierrez NR, Shoghi A, Rosander A, Pazargadi A, Ormiston CK, Wang X, Sui J, Hou Z, Fleischer JG, Golshan S, Taub PR, Panda S. Feasibility of time-restricted eating and impacts on cardiometabolic health in 24-h shift workers: The Healthy Heroes randomized control trial. Cell Metab. 2022 Oct 4;34(10):1442-1456.e7. doi: 10.1016/j.cmet.2022.08.018. PMID 36198291
- [Derived] Manoogian ENC, Zadourian A, Lo HC, Gutierrez NR, Shoghi A, Rosander A, Pazargadi A, Wang X, Fleischer JG, Golshan S, Taub PR, Panda S. Protocol for a randomised controlled trial on the feasibility and effects of 10-hour time-restricted eating on cardiometabolic disease risk among career firefighters doing 24-hour shift work: the Healthy Heroes Study. BMJ Open. 2021 Jun 16;11(6):e045537. doi: 10.1136/bmjopen-2020-045537. PMID 34135038